CLINICAL TRIAL: NCT03736837
Title: A Multi-center, One-arm Clinical Study of Anlotinib Combined With Icotinib as the First-line Treatment in Patients With EGFR Mutation-positive Advanced NSCLC. The Trial Aims to Evaluate the Efficacy and Safety of This Treatment.
Brief Title: Study of Anlotinib Combined With Icotinib as the First-line Treatment in Patients With EGFR Mutation-positive NSCLC
Acronym: ALTER-L004
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L004
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2018-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: sensitive EGFR mutations; anlotinib; icotinib; first line; cancer; non-squamous NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — anlotinib; icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Plus Icotinib (Experimental): Anlotinib 12 mg once a day from day 1 to 14 of a 21-day cycle. Icotinib 125mg p.o, tid. It should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent.
  Interventions: Drug: Anlotinib Plus Icotinib

INTERVENTIONS:
Drug: Anlotinib Plus Icotinib — Anlotinib：12mg/capsule, take once when limosis in the morning. If patients suffer from AEs, they can get declined dosage (10mg or 8mg).
  Icotinib：125 mg/tablet，three times a day，fasting or serving with food. It should be continued until disease progression or intolerable toxicity or patients withdraw of consent.
  Other Names: A+T

SUMMARY:
Evaluate the efficacy and safety of Anlotinib plus Icotinib as the first-line treatment in patients with sensitive EGFR mutations advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
Anlotinib Hydrochloride is a kind of innovative medicines approved by State Food and Drug Administration（CFDA:2011L00661） which was developed by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR1、VEGFR2、VEGFR3、FGFR1/2/3、PDGFRa/β c-Kit and MET.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. 18-75years，ECOG PS：0-2，Life expectancy of more than 3 months，with measurable lesion ( RECIST1.1)
3. Histologically or cytologically confirmed, locally advanced and/or metastatic IIIB, IIIC or IV non-squamous NSCLC or recurrent non-squamous NSCLC（according to the 8th Edition of the AJCC Staging system）with EGFR 19 del and/or 21 L858R gene mutation
4. Has not received chemotherapy or other targeted therapies；For recurrent disease, adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant chemotherapy may be accepted, but recurrence occurs after ≥6 months from stopping treatment.
5. ≥1 target lesion that has not received radiotherapy in the past 3 months and can be accurately measured in at least 1 direction；Previously received radiation therapy, but the radiotherapy area must be <25% of the bone marrow area, and radiation therapy must have closed for at least≥4 weeks at the time of enrollment;
6. Main organs function is normal
7. Patients of brain metastases with asymptomatic or mild symptoms can be enrolled
8. The woman patients of childbearing age must agree to take contraceptive methods during the research and within another 8 weeks after treatment. Pregnancy test (blood serum test or urine) should be done within 7 days before the research and the result should be negative.The man patients who must agree to take contraceptive methods during the research and within another 8 weeks after treatment.

Exclusion Criteria:

1. Squamous cell carcinoma (including adenosquamous carcinoma); Small Cell Lung Cancer (including small cell cancer and other kinds of cancer mixed with non-small cell cancer)
2. ALK-positive NSCLC
3. Central Lung tumors that Imaging (CT or MRI) shows tumor lesions invade local large blood vessels; or with significant pulmonary cavum or necrotizing
4. Patients with obvious brain metastases, cancerous meningitis, spinal cord compression, or with brain or pia mater disease. (patient with brain metastases who have completed treatment 14 days before and the symptoms are stable can be Enrolled, also should have no cerebral hemorrhage symptoms confirmed by brain MRI, CT or venography evaluation
5. The patient is participating in other clinical studies or Participated in other anti-tumor drug clinical trials within 4 weeks before enrollment
6. With other active malignancies that require simultaneous treatment
7. Has a history of malignant tumors. Except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone curative treatment and have no disease recurrence within 5 years after the start of treatment
8. Patients with adverse reactions derived from previous therapies (excluding hair loss), which is over level 1 in CTC AE (4.0)
9. abnormal blood coagulation (INR>1.5 or PT > ULN + 4s or APTT > 1.5 ULN), with bleeding tendency or receiving thrombolytic or anticoagulant therapy
10. renal insufficiency: urinary protein ≥ ++, or 24-hour urine protein ≥ 1.0g;
11. The effect of surgery or trauma has been eliminated for less than 14 days before enrollment
12. Severe acute or chronic infections requiring systemic treatment
13. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias
14. Patients with peripheral neuropathy which is over level 2 in CTC AE (4.0), except for trauma
15. respiratory syndrome (dyspnea≥CTC AE 2), severe pleural effusion, ascites, pericardial effusion
16. Long-term unhealed wounds or fractures
17. Decompensated diabetes or other ailments treated with high doses of glucocorticoids
18. with kinds of factors which affect oral medicine (e.g. failing to swallow, gastrointestinal tract getting resected, chronic diarrhea and ileus)
19. hemoptysis (daily hemoptysis>50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency
20. Thrombosis events occurring within 12 months prior to enrollment
21. Planned to get systemic anti-tumor therapy during this study；EF-RT was performed within 4 weeks before enrollment or limited field radiotherapy within 2 weeks before grouping
22. Hypertension (systolic blood pressure≥140 mmHg or diastolic blood pressure≥90 mmHg) that is still uncontrollable using two or more combination therapies
23. History of psychotropic substance abuse and inability to quit or have mental disorders
24. HIV test positive history or AIDS; untreated active hepatitis; combined with hepatitis B and hepatitis C co-infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
PFS（Progress free survival） | each 42 days up to PD or death (up to 24 months)
  The PFS time is defined as time from enrollment to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of : "death", "last tumor assessment", "last follow up date" or "last date in drug log"

SECONDARY OUTCOMES:
OS（Overall Survival） | From enrollment until death (up to 24 months)
  OS was defined as time from date of enrollment to date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.
ORR（Objective Response Rate） | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule Plus Icotinib Hydrochloric Tablet by enhanced CT/MRI scan every two cycles. Objective Response Rate (ORR) is defined as participants who had complete response (CR) or partial response(PR) divided by the total number of patients.
DCR（Disease Control Rate） | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule Plus Icotinib Hydrochloric Tablet by enhanced CT/MRI scan every two cycles. Disease Control Rate (DCR) defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease).
Adverse Events | Until 30 day safety follow-up visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, Doctor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (5):
- China (5):
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - Neimenggu Autonomous Region People's Hospital, Hohhot, Neimenggu
  - Neimenggu Medical University Affiliated Hospital, Hohhot, Neimenggu
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
De-identified individal participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requesdtors will be required to sign a Data Access Agreement.
URL: http://www.cttq.com/

REFERENCES:
- [Result] Seto T, Kato T, Nishio M, Goto K, Atagi S, Hosomi Y, Yamamoto N, Hida T, Maemondo M, Nakagawa K, Nagase S, Okamoto I, Yamanaka T, Tajima K, Harada R, Fukuoka M, Yamamoto N. Erlotinib alone or with bevacizumab as first-line therapy in patients with advanced non-squamous non-small-cell lung cancer harbouring EGFR mutations (JO25567): an open-label, randomised, multicentre, phase 2 study. Lancet Oncol. 2014 Oct;15(11):1236-44. doi: 10.1016/S1470-2045(14)70381-X. Epub 2014 Aug 27. PMID 25175099
- [Derived] Zhang L, Wang L, Wang J, Chen J, Meng Z, Liu Z, Jiang X, Wang X, Huang C, Chen P, Liang Y, Jiang R, Wang J, Zhong D, Shang Y, Zhang Y, Zhang C, Huang D. Anlotinib plus icotinib as a potential treatment option for EGFR-mutated advanced non-squamous non-small cell lung cancer with concurrent mutations: final analysis of the prospective phase 2, multicenter ALTER-L004 study. Mol Cancer. 2023 Aug 5;22(1):124. doi: 10.1186/s12943-023-01823-w. PMID 37543587
- See also: Erlotinib Plus Bevacizumab Phase ll Study in Patients with Advanced Non-small-Cell Lung Cancer (JO25567): Updated Safety Results — http://doi.org/10.1007/s40264-017-0596-0
- See also: NEJ026: Phase III study comparing bevacizumab plus erlotinib to erlotinib in patients with untreated NSCLC harboring activating EGFR mutations — http://doi.org/10.1093/annonc/mdw383.86
- See also: Phase III study comparing bevacizumab plus erlotinib (BE) to erlotinib (E) in patients (pts) with untreated NSCLC harboring EGFR mutations: NEJ026 — https://doi.org/10.1093/annonc/mdy292.063